CLINICAL TRIAL: NCT05316480
Title: Preliminary Exploration of Therapeutic Efficacy of Nimotuzumab in EGFR Highly Expressed Pancreatic Neuroendocrine Neoplasms
Brief Title: Nimotuzumab in EGFR Highly Expressed Pancreatic Neuroendocrine Neoplasms
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-1
Record Dates: First submitted 2022-03-28; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Neuroendocrine Neoplasm
Keywords: EGFR; nimotuzumab; Pancreatic Neuroendocrine Neoplasm
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab (Experimental): nimotuzumab 200mg/week
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — nimotuzumab 200mg/week

SUMMARY:
The phase II study is performed to assess the efficacy and safety of Nimotuzumab in patients with stage IV pancreatic neuroendocrine neoplasms and EGFR overexpression.

DETAILED DESCRIPTION:
Nimotuzumab (hR3) is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with various types of cancer with EGFR overexpression. The phase II study is performed to assess the efficacy and safety of Nimotuzumab in patients with stage IV pancreatic neuroendocrine neoplasms and EGFR overexpression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven diagnosis of pancreatic neuroendocrine tumors (pNET) with well and moderately differentiated with evidence of unresectable disease or metastatic disease. Locally advanced disease must not be amendable to resection or radiation therapy with curative intent.
2. Overexpression of EGFR in tumor tissue sample from tumor biopsy or prior primary tumor resection. Therefore availability of paraffin-embedding tumor tissue sample is needed.
3. Documented progression of the disease by CT scan, MRI, or Octreoscan within 12 months prior to baseline.
4. Measurable disease as per RECIST. Measurable lesions that have been previously radiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy.
5. Male or female, 18 years of age or older.
6. ECOG performance status less than 2.
7. Life expectancy greater than 12 weeks.
8. The definitions of minimum adequacy for organ function required prior to study entry are as follows.

   Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) < 2.5 x upper limit of normal (ULN), or AST and ALT < 5 x ULN if liver function abnormalities are due to underlying malignancy Total serum bilirubin < 1.5 x ULN Serum albumin > 3.0 g/dL Absolute neutrophil count (ANC) > 1500/L Hemoglobin > 9.0 g/dL Creatinin clearance < 40 mL/min
9. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Active second primary malignancy or history of second primary malignancy.
2. Current treatment on another clinical trial.
3. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus.
4. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to randomization.
5. Pathological confirmed to be poor differentiated tumor of pancreatic neuroendocrine neoplasms.
6. Patients who are unwilling or unable to comply with study procedures.
7. Prior targeted treatment on EGFR.
8. Low expression or absence of EGFR in tumor tissue sample from tumor biopsy or prior primary tumor resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Baseline to 6 months
  Overall Response rate was defined as the proportion of patients with a best overall response of complete response or partial response, based on investigator's assessment as per RECIST criteria version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Baseline to 6 months
  Disease control rate was defined as the proportion of patients with a best overall response of Complete Response, Partial response, or Stable disease, based on the investigator's assessment per RECIST version 1.1.
Progression free survival (PFS) | Patients will be followed until disease progression, estimating around 12months
Overall survival (OS) | Patients will be followed until disease progression, estimating around 12months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China